CLINICAL TRIAL: NCT03864653
Title: Brief Depression Intervention to Optimize Intensive Outpatient Methamphetamine Treatment Among Gay and Bisexual Men Who Have Sex With Men
Brief Title: Depression Intervention Among Gay and Bisexual Men Receiving Treatment for Methamphetamine Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20182627; P30MH058107 (NIH)
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: HIV/AIDS; Methamphetamine Abuse; Depression
Keywords: MSM; PrEP; ART; Sexual Risk Behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Intervention Model Description: Participants who have already enrolled in the methamphetamine outpatient treatment program, and who are still within their first two weeks of treatment, will be offered the chance to co-enroll in a low-intensity depression intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MoodGym (Other): Non-randomized single-arm intervention; eligible persons are newly enrolled methamphetamine use treatment service program (i.e., "Getting Off") participants who will be invited to participate in the study during their enrollment, and can enroll in the study at any time during their first two weeks of program participation. Participants who enroll will take the preexisting, low-intensity MoodGym intervention.
  Interventions: Behavioral: MoodGym

INTERVENTIONS:
Behavioral: MoodGym — MoodGym is a preexisting Internet-based CBT program that uses interactive content and character-driven narratives to help alleviate symptoms of depression and comorbid anxiety. The program also aims to improve the individual's functioning by promoting the development of skills and strategies to manage depression.
  MoodGym consists of an introduction module, five structured intervention modules, and a workbook of assessments. Each MoodGym session takes place entirely on an Internet-connected tablet while in the physical co-presence of a Study Counselor, who can answer questions should they arise. Each session takes approximately one hour to complete.

SUMMARY:
This study is a single-arm, non-randomized pilot study. Eligible participants are newly enrolled participants in an outpatient methamphetamine treatment program, and study activities will take place contemporaneously with participation in the service program. During the first two weeks of the treatment program, participants will be offered the chance to enroll in a low-intensity, internet-based depression intervention called MoodGym. Participants that agree to enroll will be offered the chance to attend up to seven MoodGym sessions at the same time they undergo outpatient methamphetamine treatment. It is hypothesized that sexual risk outcomes, as well as medication adherence (e.g., PrEP/PEP; ART) outcomes will be optimized for participants who enroll to receive the MoodGym intervention content.

DETAILED DESCRIPTION:
Participants will be recruited from the Getting Off service program at Friends Community Center. Program participants will be invited to participate in the study at the time that they enroll in the program, and may enroll in the study at any time during their first or second week of program participation. Getting Off program staff will inform new participants about the research study. If the potential participant is interested in learning more about the study he will be directed to meet with the Study Counselor. Both the program staff and the SC will emphasize that participation in this study is voluntary and that participation in the program is not dependent on participation in this study. Interested participants will meet with the in a private room, then read the consent form, have questions answered by the, and sign the consent form if they wish to participate.

All in-person contact (recruitment, screening, consenting, MoodGym sessions, and administration of follow-up interviews) with participants will take place in a private room with a closed door at Friends Community Center. Any telephone calls made to participants during the course of the study will be made from a private office with a closed door, so the phone conversation cannot be heard.

MoodGym is an Internet-based CBT program that uses fun, engaging, interactive content, alongside character-driven narratives, to help alleviate symptoms of depression and comorbid anxiety. The program also aims to improve the individual's functioning by promoting the development of skills and strategies to manage depression.

MoodGym consists of an introduction module, five structured intervention modules, and a workbook of assessments.

1. Getting Started

   a. An introduction to MoodGym, including CBT, the different characters and structure of the intervention content, and baseline mental health quizzes (e.g., depression, anxiety) that are scored in real time to help the participant understand their current level of mental health symptoms. This will be done during the first MoodGym session, given its brevity and relationship to the first module.
2. Feelings Module

   a. Understanding emotions, mood, and physical reactions of depression and anxiety, as well as the impact of your perspective on your personal feelings. Demonstrates links between events, thoughts, feelings, and behaviors.
3. Thoughts Module

   a. Addresses unwelcome, unhealthy, or intrusive thoughts, and demonstrates how some thoughts can help you overcome mental health symptoms. Discusses how to improve self-esteem by changing thought patterns.
4. Unwarping Module

   a. Introduces the idea of "warpy" thoughts, including false impressions that one must be perfect, that one can control all things, or that one is worthless if they are criticized.
5. Destressing Module

   1. Discusses means and strategies to reduce stress, which can have important impacts on depression and anxiety symptoms, and mental health more generally.
6. Relationships Module

   a. Discusses how relationships can both benefit or worsen one's mental health, and how to monitor and maintain healthy relationships.
7. Workbook a. Contains all quizzes and tests the participant encounters during each of the above sessions. If a participant would like to retest themselves on some dimension (e.g., depression, anxiety, warpy thoughts), they can revisit the assessment in the Workbook section, and receive an updated score in real time.

Each MoodGym session will last up to one hour and will begin with the brief CESD-R assessment, administered by the Study Counselor via the same computer as the MoodGym intervention, followed by one of the five online modules, which are self-contained and guide the participant through all intervention content. Online modules include quizzes, videos, characters, interactive activities, informational content, personal stories, workbook activities, and content summaries. Sessions can also include interactions with the Study Counselor, as much or as little as the participant chooses to initiate, including supportive feedback, guidance, help, and encouragement on activities.

The SC will monitor participant attendance and conduct a phone call to any participant who does not attend a session for two consecutive weeks.

Participants will be assessed one final time, receiving both the ART and PrEP Uptake and Adherence form and the CESD-R, at 90 days post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled within the "Getting Off" (AKA, "Friends Getting Off") outpatient methamphetamine treatment program at Friends Community Center, Los Angeles, CA, USA.
* and; within two weeks of initial enrollment into the "Getting Off" program.

Exclusion Criteria:

* Not currently enrolled within the "Getting Off" program.
* or; more than two weeks post-enrollment in the "Getting Off" program.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse B Fletcher, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Community Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data with other researchers.

REFERENCES:
- See also: MoodGym Intervention — http://moodgym.com.au/
- See also: Getting Off Treatment Manual — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=10&ved=2ahUKEwjZ4v7q3OHgAhXW7Z4KHQs6DiQQFjAJegQIAhAC&url=http%3A%2F%2Fwww.uclaisap.org%2Fassets%2Fdocuments%2FShoptawetal_2005_tx%2520manual.pdf&usg=AOvVaw1hngtTYTH3I4gME5GHYoo4

RESULTS

PARTICIPANT FLOW:
Groups:
- MoodGym: Non-randomized single-arm intervention; eligible persons are newly enrolled methamphetamine use treatment service program (i.e., "Getting Off") participants who will invited to participate in the study during their enrollment, and can enroll in the study at any time during their first two weeks of program participation. Participants who enroll will take the preexisting, low-intensity MoodGym intervention.
  MoodGym: MoodGym is a preexisting Internet-based CBT program that uses interactive content and character-driven narratives to help alleviate symptoms of depression and comorbid anxiety. The program also aims to improve the individual's functioning by promoting the development of skills and strategies to manage depression.
  MoodGym consists of an introduction module, five structured intervention modules, and a workbook of assessments. Each MoodGym session takes place entirely on an Internet-connected tablet while in the physical co-presence of a Study Counselor, who can answe
Period: Overall Study
Arm/Group | MoodGym
Started | 39
Completed | 38
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MoodGym
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.87 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Black | 4
  Latinx | 19
  Multiracial/Multiethnic/Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 38
Tenure of Heavy Methamphetamine Use [Mean (Standard Deviation); unit: years] — Participants were asked "How long have you been using methamphetamine heavily?", and responses were measured in "years."
  years | 5.11 (5.41)
Methamphetamine Use [Mean (Standard Deviation); unit: days] — Participants were asked "How many days in the past 30 days have you used methamphetamine?"
  days | 8.11 (9.23)

OUTCOME MEASURES:

1. Primary Outcome: Depression Symptoms Over Time
Description: Depression symptoms are measured using the Center for Epidemiologic Studies Depression Scale (Revised; CESD-R) to begin each MoodGym session. The CESD-R consists of 20 items, each of which is a statement that participants are asked to endorse on a five-point scale from "not at all or less than one day in the last week" to "nearly every day for two weeks." Scores range from 0 thru 80, with higher scores indicating greater depression symptomology. The outcome measure described below indicates the average change in CESD-R scores for each MoodGym session attended.
Time Frame: Last Two Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | MoodGym
Number analyzed (Participants) | 38
Units on a Scale | -0.062 [-0.095 to -0.030]

2. Primary Outcome: HIV-Related Medication Adherence
Description: A participant's self-reported adherence to ART (HIV-positive participants) or PrEP (HIV-negative participants) will be assessed via a short questionnaire. HIV-positive participants are asked if they are on an antiretroviral regimen (i.e., ART), and if so, when they began the regimen and their recent adherence patterns. HIV-negative participants are asked if they know what pre-exposure prophylaxis (PrEP) is, whether they are on PrEP, and if so, when they began the regimen.
Time Frame: Last 90 Days
Population: HIV-Positive Study Participants who reported on their ART medication adherence at 90-day follow-up (zero HIV-negative participants enrolled who reported being on PrEP).
Measure: Mean (Standard Deviation); unit: doses missed
Arm/Group | MoodGym
Number analyzed (Participants) | 9
doses missed | 4.78 (3.87)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | MoodGym
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 2/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MoodGym (N=39)
Blood Clot (Blood and lymphatic system disorders) | 1 (1) — Mood Gym Participant was hospitalized in May 2019 due to a blood clot.
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — Mood Gym Participant was hospitalized in June 2019 for breakout of cellulitis.

LIMITATIONS AND CAVEATS:
COVID-19 pandemic travel restrictions reduced ability to conduct timely follow-up in the final months of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03864653/Prot_SAP_000.pdf